CLINICAL TRIAL: NCT06284967
Title: A Prospective Study On Association Of Serum Vitamin D Level With Isthmic Spondylolysis In Adult Population
Brief Title: Association Of Serum Vitamin D Level With Isthmic Spondylolysis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Emad Zakaria Nasif, Principal investigator, Assiut University
Other Study IDs: Vitamin D In Spondylolysis
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Spondylolysis
MeSH Terms: conditions — Spondylolysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Adults aged 20 - 45 years with symptomatic isthmic spondylolysis
- Controls: Matched population without spondylolysis indicated for plain x-ray and CT lumbo-sacral spine. These will be recruited mainly from the Trauma Unit. This will not add any non-indicated radiation exposure to healthy individuals

SUMMARY:
The aim of this study is to compare vitamin D level between young adults with isthmic spondylolysis and a matched healthy control group.

DETAILED DESCRIPTION:
Deficiency of 25-hydroxy vitamin D has been of recent interest , and its high prevalence has been confirmed across all age groups in many cross sectional studies, particularly in developing countries and in the Middle East and Northern Africa Region . The formation and maintenance of a structurally stiff and resilient skeleton is dependent upon vitamin D's role in absorption of calcium from the gut and in normal bone metabolism thereafter. Failure of adequate mineral accretion reduces normal bone turnover and may result in rickets, osteomalacia, and osteoporosis later in life . Several risk factors for hypovitaminosis D have been described in the literature, including nutrition, little exposure to ultraviolet light, darker skin pigmentation, and lack of physical activity .

Lumbar isthmic spondylolysis is a stress fracture of the pars interarticularis, which is generally considered a disease of adolescents and young adults .

The exact prevalence of spondylolysis in our region is not exactly known, but the general impression among spine surgeons is that it is much higher than the 3-6% prevalence reported for the Caucasian population .

Spondylolysis commonly affects children and young adults . The exact etiology of this fatigue fracture of the pars interarticularis is still not well understood . The most probable mechanism of lumbar spondylolysis is multifactoral with a stress fracture occurring through a weak or dysplastic pars interarticularis. The likely initiating event occurs when the patient engages in repeated extension and/or axial rotation maneuvers .

Vitamin D deficiency may be a predisposing factor to weak bone and subsequent fractures . Despite abundant sunshine, hypovitaminosis D is very common in the Middle East Region and several cross- sectional studies in Egypt , Iran , Tunisia , Jordan , United Arab Emirates, and other Gulf countries have been reported. Symptomatic spondylolysis is indicated for surgical intervention.

Currently, children and adolescents with spondylolysis are treated with pars reconstruction techniques. Adults with symptomatic isthmic spondylolysis or with large defects are treated with spinal fusion.

The hypothesis of this study is that hypovitaminosis D predisposes to weakness of the pars interarticularis and subsequently is a risk factor for developing isthmic spondylolysis. Given the common incidence of hypovitaminosis D in Egyptian population and the negative impact of spondylolysis on the young active age group, this study would have important implications regarding prophylactic vitamin D supplementation as well as the prevention of spondylolysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Adults aged 20 - 45 years with symptomatic isthmic spondylolysis
* Controls: Matched population without spondylolysis indicated for plain x-ray and CT lumbo-sacral spine. These will be recruited mainly from the Trauma Unit. This will not add any non-indicated radiation exposure to healthy individuals

Exclusion Criteria:

* Traumatic spondylolysis
* Pregnant women
* Significant co-morbidities (renal or hepatic diseases, malignancy, malabsorption syndrome, musculoskeletal diseases, steroid therapy)
* Metabolic diseases affecting vitamin D and Calcium metabolism (e.g. hyperparathyroidism)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Detailed history taking (including dietary calcium and vitamin D intakes, Exposure to sun, and Clothing habits)
  * Clinical examination
  * Imaging: plain x-ray and CT scan
  * Laboratory: Free serum calcium, alkaline phosphatase and 25-OH vitamin D
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean serum vitamin D in both groups. | Baseline
  Patients will be classified, according to the Endocrine Society guidelines for 2011, into vitamin D deficient if serum 25 is ≤20 ng/dl, vitamin D insufficient if it is 21-29 ng/dl and vitamin D sufficient if it is ≥30 ng/dl [8].

SECONDARY OUTCOMES:
Mean serum calcium level | Baseline
  Mean serum Calcium level in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shawky Abdelgawaad, Professor, Study Director — Assiut University; Mahmoud Fouad Ibrahim, Doctor, Principal Investigator — Assiut University

REFERENCES:
- [Background] McClellan JW 3rd, Vernon BA, White MA, Stamm S, Ryschon KL. Should 25-hydroxyvitamin D and bone density using DXA be tested in adolescents with lumbar stress fractures of the pars interarticularis? J Spinal Disord Tech. 2012 Dec;25(8):426-8. doi: 10.1097/BSD.0b013e31823f324f. PMID 22134731
- [Background] Chakhtoura M, Rahme M, Chamoun N, El-Hajj Fuleihan G. Vitamin D in the Middle East and North Africa. Bone Rep. 2018 Mar 17;8:135-146. doi: 10.1016/j.bonr.2018.03.004. eCollection 2018 Jun. PMID 29955632
- [Background] Bassil D, Rahme M, Hoteit M, Fuleihan Gel-H. Hypovitaminosis D in the Middle East and North Africa: Prevalence, risk factors and impact on outcomes. Dermatoendocrinol. 2013 Apr 1;5(2):274-98. doi: 10.4161/derm.25111. PMID 24194968
- [Background] Melamed ML, Kumar J. Low levels of 25-hydroxyvitamin D in the pediatric populations: prevalence and clinical outcomes. Ped Health. 2010 Feb;4(1):89-97. doi: 10.2217/phe.09.72. PMID 20490283
- [Background] Prentice A, Goldberg GR, Schoenmakers I. Vitamin D across the lifecycle: physiology and biomarkers. Am J Clin Nutr. 2008 Aug;88(2):500S-506S. doi: 10.1093/ajcn/88.2.500S. PMID 18689390
- [Background] Kalkwarf HJ, Zemel BS, Gilsanz V, Lappe JM, Horlick M, Oberfield S, Mahboubi S, Fan B, Frederick MM, Winer K, Shepherd JA. The bone mineral density in childhood study: bone mineral content and density according to age, sex, and race. J Clin Endocrinol Metab. 2007 Jun;92(6):2087-99. doi: 10.1210/jc.2006-2553. Epub 2007 Feb 20. PMID 17311856
- [Background] Holick MF. Vitamin D: importance in the prevention of cancers, type 1 diabetes, heart disease, and osteoporosis. Am J Clin Nutr. 2004 Mar;79(3):362-71. doi: 10.1093/ajcn/79.3.362. PMID 14985208
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Holick MF. Vitamin D: a d-lightful solution for health. J Investig Med. 2011 Aug;59(6):872-80. doi: 10.2310/JIM.0b013e318214ea2d. PMID 21415774
- [Background] Fredrickson BE, Baker D, McHolick WJ, Yuan HA, Lubicky JP. The natural history of spondylolysis and spondylolisthesis. J Bone Joint Surg Am. 1984 Jun;66(5):699-707. PMID 6373773
- [Background] Virta L, Ronnemaa T, Osterman K, Aalto T, Laakso M. Prevalence of isthmic lumbar spondylolisthesis in middle-aged subjects from eastern and western Finland. J Clin Epidemiol. 1992 Aug;45(8):917-22. doi: 10.1016/0895-4356(92)90075-x. PMID 1624974
- [Background] Albanese M, Pizzutillo PD. Family study of spondylolysis and spondylolisthesis. J Pediatr Orthop. 1982;2(5):496-9. doi: 10.1097/01241398-198212000-00006. PMID 6761366
- [Background] Saraste H. Long-term clinical and radiological follow-up of spondylolysis and spondylolisthesis. J Pediatr Orthop. 1987 Nov-Dec;7(6):631-8. PMID 2963019
- [Background] Lawrence KJ, Elser T, Stromberg R. Lumbar spondylolysis in the adolescent athlete. Phys Ther Sport. 2016 Jul;20:56-60. doi: 10.1016/j.ptsp.2016.04.003. Epub 2016 Apr 13. PMID 27234265
- [Background] Farouk O, Mahran DG, Said HG, Alaa MM, Eisa AA, Said GZ, Rashed H, Ez-Eldeen A. Hypovitaminosis D Among Patients Admitted With Hip Fracture to a Level-1 Trauma Center in the Sunny Upper Egypt: Prevalence and Associated Correlates. Geriatr Orthop Surg Rehabil. 2016 Sep;7(3):148-52. doi: 10.1177/2151458516655436. Epub 2016 Jun 22. PMID 27551573
- [Background] Botros RM, Sabry IM, Abdelbaky RS, Eid YM, Nasr MS, Hendawy LM. Vitamin D deficiency among healthy Egyptian females. Endocrinol Nutr. 2015 Aug-Sep;62(7):314-21. doi: 10.1016/j.endonu.2015.03.010. Epub 2015 Jun 10. English, Spanish. PMID 26070223
- [Background] Hashemipour S, Larijani B, Adibi H, Javadi E, Sedaghat M, Pajouhi M, Soltani A, Shafaei AR, Hamidi Z, Fard AR, Hossein-Nezhad A, Booya F. Vitamin D deficiency and causative factors in the population of Tehran. BMC Public Health. 2004 Aug 25;4:38. doi: 10.1186/1471-2458-4-38. PMID 15327695
- [Background] Meddeb N, Sahli H, Chahed M, Abdelmoula J, Feki M, Salah H, Frini S, Kaabachi N, Belkahia Ch, Mbazaa R, Zouari B, Sellami S. Vitamin D deficiency in Tunisia. Osteoporos Int. 2005 Feb;16(2):180-3. doi: 10.1007/s00198-004-1658-6. Epub 2004 Jun 10. PMID 15197539
- [Background] Mishal AA. Effects of different dress styles on vitamin D levels in healthy young Jordanian women. Osteoporos Int. 2001;12(11):931-5. doi: 10.1007/s001980170021. PMID 11804019
- [Background] Lips P, Hosking D, Lippuner K, Norquist JM, Wehren L, Maalouf G, Ragi-Eis S, Chandler J. The prevalence of vitamin D inadequacy amongst women with osteoporosis: an international epidemiological investigation. J Intern Med. 2006 Sep;260(3):245-54. doi: 10.1111/j.1365-2796.2006.01685.x. PMID 16918822
- [Background] Saadi HF, Nagelkerke N, Benedict S, Qazaq HS, Zilahi E, Mohamadiyeh MK, Al-Suhaili AI. Predictors and relationships of serum 25 hydroxyvitamin D concentration with bone turnover markers, bone mineral density, and vitamin D receptor genotype in Emirati women. Bone. 2006 Nov;39(5):1136-1143. doi: 10.1016/j.bone.2006.05.010. Epub 2006 Jun 30. PMID 16814623
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343